CLINICAL TRIAL: NCT04880863
Title: Phase 2a Open-Label, Multicenter Trial of Naptumomab Estafenatox (NAP) in Combination With Docetaxel Following Obinutuzumab Pretreatment in Subjects With Checkpoint Inhibitor Pretreated Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: NAP in Combination With Docetaxel Following Obinutuzumab Pretreatment in Subjects With Checkpoint Inhibitor Pretreated Advanced or Metastatic NSCLC
Acronym: NT-NAP-102-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeoTX Therapeutics Ltd. (Industry)
Collaborators: Translational Drug Development (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NT-NAP-102-1
Record Dates: First submitted 2021-05-03; First posted 2021-05-11 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Advanced; Metastatic; Non small cell lung cancer; EGFR; ALK; Docetaxel; Naptumomab estafenatox; Obinutuzumab; NAP
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — naptumomab estafenatox; Docetaxel; obinutuzumab

STUDY DESIGN:
Intervention Model Description: Subjects receive obinutuzumab, 1,000 mg, administered by IV infusion on Days -13 and -12 of the first treatment cycle in order to reduce the titer of anti-drug antibodies to NAP. NAP is administered by IV bolus on Days 1 - 4 of treatment cycles 1-6, followed by docetaxel on Day 5. Treatment cycles with the combination NAP/docetaxel are of 21 days in duration. Starting cycle 7, NAP at a higher dose is administered on Day 1 and docetaxel on Day 2, in 21 days treatment cycles. Once NAP is given as monotherapy and not earlier than C7, cycles are of 28 days of duration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NAP in combination with docetaxel following obinutuzumab pretreatment (Experimental): Subjects receive obinutuzumab, 1,000 mg, administered by IV infusion on Days -13 and -12 of the first treatment cycle in order to reduce the titer of anti-drug antibodies to NAP. NAP is administered by IV bolus on Days 1 - 4 of treatment cycles 1-6, followed by docetaxel on Day 5. Treatment cycles with the combination NAP/docetaxel are of 21 days in duration. Starting cycle 7, NAP at a higher dose is administered on Day 1 and docetaxel on Day 2, in 21 days treatment cycles. Once NAP is given as monotherapy and not earlier than C7, cycles are of 28 days of duration.
  Interventions: Drug: NAP (Naptumomab estafenatox); Drug: Docetaxel; Drug: Obinutuzumab

INTERVENTIONS:
Drug: NAP (Naptumomab estafenatox) — Naptumomab estafenatox (NAP; ABR-217620) is a recombinant fusion protein consisting of a chimeric staphylococcal enterotoxin A/E (SEA/SEE) superantigen with several additional substitutions that are linked to a Fab moiety recognizing a tumor-associated glycoprotein, 5T4. NAP is administered at a dose of 10 μg/kg/day by IV bolus on Days 1 - 4 of treatment cycles 1-6. Starting cycle 7, NAP at a higher dose of 15 μg/kg is administered on Day 1.
  Other Names: ABR-217620; Anyara
Drug: Docetaxel — Docetaxel is administered in combination with the study drug, NAP, on Day 5 of the treatment cycles 1-6. Starting cycle 7, Docetaxel is administered in combination with the study drug, NAP, on Day 2.
  Other Names: Taxotere
Drug: Obinutuzumab — Obinutuzumab is administered as pre-medication on Day -13 and -12 of the first treatment cycle.
  Other Names: Gazyva

SUMMARY:
Phase 2a Open-Label, Multicenter Trial of Naptumomab Estafenatox (NAP), following Obinutuzumab Pretreatment, on Days -13 and -12. NAP will be administered on Days 1-4 of treatment cycles 1-6, followed by docetaxel on Day 5. Starting cycle 7, NAP at a higher dose will be administered on Day 1 only and docetaxel on Day 2, in 21 days treatment cycles. When NAP is administered as monotherapy and not earlier than cycle 7, NAP will be administered on Day 1 only and cycles will be of 28 days treatment cycle.

DETAILED DESCRIPTION:
Patients must have received at least 1 and no more than 2 prior systemic regimens for the treatment of advanced/metastatic NSCLC. Patients were required to have progressed following treatment with both platinum-based chemotherapy and an anti-PD-(L)1 antibody administered either sequentially or concurrently. Entry into this trial was restricted to patients with incurable disease, including those whose disease had relapsed within 6 months after chemoradiotherapy for Stage III disease. Patients were to have available archival or fresh tissue collected for the retrospective determination of tumoral 5T4 levels.

ELIGIBILITY:
Main Inclusion Criteria:

1. Subjects must be at least 18 years of age
2. Subjects must have histologically and/or cytologically confirmed NSCLC
3. Subjects must have incurable (advanced or metastatic) disease at the time of enrolment
4. Subjects must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
5. Subjects must provide signed informed consent prior to any study specific procedures that are not part of standard medical care.
6. Subjects must have measurable neoplastic disease based on the iRECIST criteria
7. Subjects must have received as least 1 and no more than 2 prior systemic regimens for the treatment of advanced/metastatic NSCLC. Patients are required to have progressed following treatment with both platinum-based chemotherapy and an anti-PD-(L)1 antibody administered either sequentially or concurrently. A prior PD-1/PD-L1 inhibitor is, however, not required if there was prior exposure to targeted therapies for a driver mutation positive tumors (e.g. EGFR or ALK inhibitors).

Main Exclusion Criteria:

1. Subjects with active infection requiring treatment within 3 days of C1D1.
2. Subjects with other active neoplastic disease requiring concurrent anti-neoplastic treatment
3. Subjects with known, suspected or documented parenchymal brain metastases unless treated with surgery and/or radiation, with the subject neurologically stable and off pharmacologic doses of systemic glucocorticoids; subjects with leptomeningeal metastases are not eligible. Patients should have completed brain radiation for at least 14 days and be off steroids.
4. Active or previously documented autoimmune or inflammatory disorders such as, but not limited to rheumatoid arthritis, systemic lupus erythematosus, uveitis, ulcerative colitis, Crohn's syndrome, Wegener's syndrome, multiple sclerosis, myasthenia gravis, scleroderma and sarcoidosis. The following are exceptions to this criterion:

   * Vitiligo or psoriasis not requiring systemic treatment (within the last 2 years)
   * Subjects with endocrinopathies (e.g. following Hashimoto syndrome) stable on hormone replacement or do not require any therapy.
5. History of primary immunodeficiency
6. Subjects with a history or prior allogeneic organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Lorber, MD, Study Director — NeoTX Therapeutics Ltd.
Locations (11):
- United States (11):
  - NeoTX - 10307, Daphne, Alabama
  - NeoTX - 10302, Scottsdale, Arizona
  - NeoTX - 10303, Tucson, Arizona
  - NeoTX - 10306, Lone Tree, Colorado
  - NeoTX - 10304, Minneapolis, Minnesota
  - NeoTX - 10100, Morristown, New Jersey
  - NeoTX - 10308, Austin, Texas
  - NeoTX - 10309, Dallas, Texas
  - NeoTX - 10312, El Paso, Texas
  - NeoTX - 10310, Tyler, Texas
  - NeoTX - 10311, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NAP in Combination With Docetaxel Following Obinutuzumab Pretreatment: Subjects will receive obinutuzumab, 1,000 mg, administered by IV infusion on Days -13 and -12 of the first treatment cycle in order to reduce the titer of anti-drug antibodies to NAP. NAP will be administered in a daily dose of 10 μg/kg by IV bolus on Days 1 - 4 of treatment cycles 1-6, followed by docetaxel, 75 mg/m2 on Day 5. Treatment cycles with the combination NAP/docetaxel will be 21 days in duration. Starting cycle 7, NAP at a higher dose of 15 μg/kg will be administered on Day 1 and docetaxel on Day 2, in 21 days treatment cycles. Once NAP is given as monotherapy and not earlier than C7, cycles will be of 28 days of duration.
  NAP (Naptumomab estafenatox): Naptumomab estafenatox (NAP; ABR-217620) is a recombinant fusion protein consisting of a chimeric staphylococcal enterotoxin A/E (SEA/SEE) superantigen with several additional substitutions that is linked to a Fab moiety recognizing a tumor-associated glycoprotein, 5T4. NAP will be administered in a dose of 10 μg/kg/day by IV bolus on Days 1 - 4 of treatment cycles 1-6. Starting cycle 7, NAP at a higher dose of 15 μg/kg will be administered on Day 1.
  Docetaxel: Docetaxel is administered in combination with the study drug, NAP, on Day 5 of the treatment cycles 1-6. Starting cycle 7, Docetaxel will be administered in combination with the study drug, NAP, on Day 2.
  Obinutuzumab: Obinutuzumab is administered as pre-medication on Day -13 and -12 of the first treatment cycle.
Period: Overall Study
Arm/Group | NAP in Combination With Docetaxel Following Obinutuzumab Pretreatment
Started | 38
Completed | 0
Not Completed | 38
Not completed — Adverse Event | 1
Not completed — Patient decision | 2
Not completed — Confirmed Disease Progression | 15
Not completed — Death | 3
Not completed — Physician Decision | 4
Not completed — Unconfirmed Disease Progression | 4
Not completed — Withdrawal by Subject | 2
Not completed — Study discontinuation by the sponsor | 4
Not completed — Progression disease identified by lumbar puncture | 1
Not completed — Not received study drug NAP | 2

BASELINE CHARACTERISTICS:
Population: A single arm trial
Groups:
- NAP in Combination With Docetaxel Following Obinutuzumab Pretreatment: Subjects received obinutuzumab, 1,000 mg, administered by IV infusion on Days -13 and -12 of the first treatment cycle in order to reduce the titer of anti-drug antibodies to NAP. NAP was administered in a daily dose of 10 μg/kg by IV bolus on Days 1 - 4 of treatment cycles 1-6, followed by docetaxel, 75 mg/m2 on Day 5. Treatment cycles with the combination NAP/docetaxel were 21 days in duration. Starting cycle 7, NAP at a higher dose of 15 μg/kg was administered on Day 1 and docetaxel on Day 2, in 21 days treatment cycles. Once NAP was given as monotherapy and not earlier than C7, cycles were of 28 days of duration.
Arm/Group | NAP in Combination With Docetaxel Following Obinutuzumab Pretreatment
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 66 [33 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 33
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) and iRECIST for target lesions and assessed by CT scans or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: From the first treatment to first CR or PR (estimated about 24 months)
Population: Efficacy Evaluable Population: patients completing at least one treatment cycle and having had an evaluable pre-treatment and one post-treatment tumor assessment (according to the iRECIST - criteria) in the absence of eligibility and compliance issues.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | NAP in Combination With Docetaxel Following Obinutuzumab Pretreatment
Number analyzed (Participants) | 32
percentage of responders | 15.6 [5.3 to 32.8]

2. Secondary Outcome: Disease Control Rate (DCR)
Description: The proportion of subjects who achieve a best response of CR, PR or SD per Response Evaluation in Solid Tumors (iRECIST).
Time Frame: From the first administration of treatment till study completion (estimated about 24 months).
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients with SD, PR, CR
Arm/Group | NAP in Combination With Docetaxel Following Obinutuzumab Pretreatment
Number analyzed (Participants) | 32
percentage of patients with SD, PR, CR | 71.9 [53.3 to 86.3]

3. Secondary Outcome: Duration of Response (DOR)
Description: Duration from first documentation of CR or PR (whichever occurs first) after the first administration of obinutuzumab pretreatment until death or progressive disease (PD)
Time Frame: estimated about 24 months.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NAP in Combination With Docetaxel Following Obinutuzumab Pretreatment
Number analyzed (Participants) | 32
months | 12.2 [1.6 to 17.7]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS per Response Evaluation in Solid Tumors (iRECIST)
Time Frame: From the first administration of treatment to the date of first documentation of disease progression, or death due to any cause, whichever occurs first (estimated about 24 months).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | NAP in Combination With Docetaxel Following Obinutuzumab Pretreatment
Number analyzed (Participants) | 32
months | 8.8 [6.1 to 15.2]

5. Secondary Outcome: Overall Survival (OS)
Description: The time from first day of study drug treatment to death for any cause
Time Frame: estimated about 24 months.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | NAP in Combination With Docetaxel Following Obinutuzumab Pretreatment
Number analyzed (Participants) | 32
months | 8.8 [6.4 to 11.7]

6. Secondary Outcome: Treatment-Emergent Adverse Events (TEAEs)
Description: Number of subjects with treatment emergent adverse events as assessed by CTCAE v5.0
Time Frame: From the first administration of obinutuzumab pretreatment till study completion (estimated about 24 months).
Population: Safety Subjects Population
Measure: Number; unit: participants
Arm/Group | NAP in Combination With Docetaxel Following Obinutuzumab Pretreatment
Number analyzed (Participants) | 38
participants
  TEAE Grade 1 or 2 | 37
  TEAEs Grade ≥3 | 34
  TEAE Related to Docetaxel Grade 1 or 2 | 28
  TEAE Related to Docetaxel Grade ≥ 3 | 27
  TEAE Related to Obinutuzumab Grade 1 or 2 | 18
  TEAE Related to Obinutuzumab Grade ≥ 3 | 6
  TEAE Related to NAP Grade 1 or 2 | 33
  TEAE Related to NAP Grade ≥ 3 | 22
  TEAE Related to NAP when given as a single agent Grade 1 or 2 | 4
  TEAE Related to NAP when given as a single agent Grade ≥ 3 | 3

ADVERSE EVENTS:
Time Frame: Treatment Emergent AEs were collected from first study drug administration till 30 days post last subject last visit, i.e. through study completion, an average of 2 years.
Arm/Group | NAP in Combination With Docetaxel Following Obinutuzumab Pretreatment
All-Cause Mortality (participants affected / at risk) | 6/38
Serious Adverse Events (participants affected / at risk) | 16/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAP in Combination With Docetaxel Following Obinutuzumab Pretreatment (N=38)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Pneumonia (Infections and infestations) | 4 (4)
Neutrophil count decreased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Sepsis (Infections and infestations) | 2 (2)
Superior vena cava syndrome (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAP in Combination With Docetaxel Following Obinutuzumab Pretreatment (N=38)
Anaemia (Blood and lymphatic system disorders) | 11 (14)
Tachycardia (Cardiac disorders) | 8 (11)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 16 (25)
Diarrhoea (Gastrointestinal disorders) | 12 (16)
Vomiting (Gastrointestinal disorders) | 11 (17)
Constipation (Gastrointestinal disorders) | 11 (14)
Abdominal pain (Gastrointestinal disorders) | 8 (13)
Abdominal pain upper (Gastrointestinal disorders) | 3 (5)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Oral pain (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 24 (43)
Chills (General disorders) | 22 (37)
Pyrexia (General disorders) | 12 (17)
Pain (General disorders) | 10 (13)
Oedema peripheral (General disorders) | 8 (11)
Asthenia (General disorders) | 4 (6)
Chest pain (General disorders) | 4 (4)
Mucosal inflammation (General disorders) | 2 (2)
Pneumonia (Infections and infestations) | 6 (8)
Urinary tract infection (Infections and infestations) | 5 (5)
COVID-19 (Infections and infestations) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 2 (4)
Sinusitis (Infections and infestations) | 2 (3)
Bronchitis (Infections and infestations) | 2 (2)
Diverticulitis (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Wound complication (Injury, poisoning and procedural complications) | 2 (2)
Neutrophil count decreased (Investigations) | 21 (32)
Weight decreased (Investigations) | 7 (8)
White blood cell count decreased (Investigations) | 5 (7)
Aspartate aminotransferase increased (Investigations) | 4 (6)
Blood creatinine increased (Investigations) | 4 (5)
Gamma-glutamyltransferase increased (Investigations) | 4 (5)
Blood alkaline phosphatase increased (Investigations) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (5)
Lymphocyte count decreased (Investigations) | 2 (3)
Platelet count decreased (Investigations) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 (17)
Decreased appetite (Metabolism and nutrition disorders) | 9 (11)
Dehydration (Metabolism and nutrition disorders) | 7 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (9)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 9 (12)
Dizziness (Nervous system disorders) | 7 (7)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (6)
Dysgeusia (Nervous system disorders) | 2 (3)
Dysaesthesia (Nervous system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 5 (5)
Anxiety (Psychiatric disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (9)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5)
Nail disorder (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Hypotension (Vascular disorders) | 13 (19)
Hypertension (Vascular disorders) | 6 (11)
Flushing (Vascular disorders) | 2 (3)
Hot flush (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study Sites or Principal Investigators shall not publish the Results or the outcomes of their individual participation in the Study, until after the completion of the Study at all participating sites and the review, analysis, and write-up of the Study by the Sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT04880863/Prot_SAP_000.pdf